CLINICAL TRIAL: NCT03570801
Title: SLIP II Registry: Spinal Laminectomy to Laminectomy With Instrumented Pedicle Screw Fusion for Lumbar Stenosis With Grade I Spondylolisthesis
Brief Title: SLIP II Registry: Spinal Laminectomy Versus Instrumented Pedicle Screw Fusion
Acronym: SLIPII
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-047
Record Dates: First submitted 2018-06-12; First posted 2018-06-27 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Lumbar Spondylolisthesis; Grade 1 Spondylolisthesis; Lumbar Spinal Stenosis; Degenerative Spondylolisthesis
Keywords: Lumbar Spondylolisthesis; Grade 1 Spondylolisthesis; Lumbar Spinal Stenosis; Degenerative Spondylolisthesis
MeSH Terms: conditions — Spondylolisthesis; Spinal Stenosis

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial with randomization ratio 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Expert Panel Review (Experimental): For patients who are randomized to receive an expert panel review, de-identified lumbar MRI (sagittal and key axial images), 36-inch standing plain radiographs (if available), and flexion and extension radiographs will be uploaded into a web-based platform and reviewed. These will be submitted for an Expert Panel Review.
  Images will be reviewed through a Spine Expert's Network, consisting of physicians involved in this study who will each offer their opinion as to which of two surgical treatment groups (decompression alone or decompression with fusion) they would choose for the patient. The results of this review will be discussed between the patient and the patient's physician. Together, they will determine the best surgical approach.
  Interventions: Other: Expert Panel Review
- No Expert Panel Review (No Intervention): For patients not receiving the expert panel review, they will discuss with their surgeon the best surgical option and proceed as they would in standard of care.

INTERVENTIONS:
Other: Expert Panel Review — There is some preliminary evidence suggesting that having a group of spinal experts review x-rays prior to treatment might provide useful information to the patient and the patients' treating physician when trying to make a decision about what type of surgery to perform.
  Arms: Expert Panel Review

SUMMARY:
The purpose of the project is to perform an RCT comparing patient satisfaction and outcome with or without the use of an expert panel. The purpose is also to create a registry to compare the effectiveness of decompression alone versus decompression with fusion for patients with degenerative grade I spondylolisthesis and symptomatic lumbar spinal stenosis. Primary analysis will focus on the patients' improvement from baseline patient-reported outcome questionnaires.

In addition, the SLIP II registry aims to (i) develop an algorithm which could identify cases in which surgical experts are likely to recommend one treatment (i.e. >80% of experts recommend one form of treatment) and (ii) develop a radiology-based machine learning algorithm that would prospectively classify patients as either 'stable' or 'unstable.'

In addition to patient reported outcomes, step counts will be collected in order to determine the correlation of step count with patient-reported outcomes (ODI and EQ-5D) and the need for re-operation.

This registry portion of the study aims to prospectively collect comparative data for these patients treated with either decompression alone or decompression with fusion.

DETAILED DESCRIPTION:
Aim: To conduct a randomized control trial comparing patient outcomes and satisfaction with or without expert panel review before making a final decision about surgery for grade I degenerative lumbar spondylolisthesis. A prospective, multi-center registry aimed at addressing important issues pertaining to outcomes from treatment for degenerative spondylolisthesis and spinal stenosis will also be generated.

Background: Surgery may be offered to patients with symptomatic lumbar stenosis with degenerative lumbar spondylolisthesis who fail nonoperative treatment measures including physical therapy and epidural steroid injections. For patients with lumbar stenosis without spondylolisthesis, a decompression alone is typical, while those patients who do have degenerative spondylolisthesis and who also have significant mechanical back pain may be offered lumbar decompression with or without fusion. These guidelines were written based upon the SPORT study, which provided the highest quality of evidence available at the time. Additional studies have show that costly interventions such as lumbar fusion may ultimately be cost-effective if they provide durable clinical benefit. Two recent publications in The New England Journal of Medicine present new evidence with conflicting results on superficial review. The Spinal Laminectomy versus Instrumented Pedicle Screw (SLIP) trial provides level I evidence for the efficacy of fusion to improve clinical outcomes and lower reoperation rates compared to a standard laminectomy and medial facetectomy over a four year time frame in patients with neurogenic claudication associated with stable single level spondylolisthesis. Conversely, the Swedish study provides level II evidence that the addition of a variety of fusion techniques does not have significant benefit in the first two years following operation compared to a variety of decompression techniques in a heterogeneous population of patients with stenosis associated with spondylolisthesis. The patient populations treated, surgical techniques used, and outcome measures assessed differed between the two studies and when taken together, underline the need to new comparative effectiveness data for patients with this problem.

Additionally, one key challenge surgeons face is whether or not to recommend a spinal fusion. Spinal fusion is expensive, assoicated with greater costs and complications, but it appears to be necessary in at least 30% of patients.3 Preliminary data suggests that when when greater than 80% of an expert panel votes for one treatment opition, either a fusion or decompression alone, and when a patient's actual treatment aligns with the expert panel recommention, the patient-reported outcomes are greater than when the surgical approach is not aligned with the expert panel.10 This data highlights an interest in developing articifical intelligence (AI) that may be able to aid in both identification and predictive tasks. Any progress in this realm would be enormously powerful from a clinical standpoint and would likely result in more efficient use of surgical appraoches and in turn, healthcare spending.

All images that are captured in the registry will be used to train convolutional neural networks (CNN). These are mathematical operations which extract patterns from image data and generalize it across many images fed into the dataset. They primarily use calculations to extract patterns which are stored as a model which will be a collection of numbers. The images stored in this registry will be used to develop algorithms to assess cases in which an expert panel is more likely to suggest one treatment over the other as well as develop an algorithm that would prospectively classify patients as either 'stable' or 'unstable.'

Plan: Before making a decision regarding which specific operation should be performed in each case, each patient will be randomized to receive an expert panel review or to not receive an expert panel review. For patients who receive an expert panel review, the patients' de-identified lumbar MRI (sagittal and key axial images), 36-inch standing plain radiographs (if available), and flexion and extension radiographs will be uploaded into a web-based platform and reviewed with plans to share the reviews with patients and their treating physicians in real time. For patients who are randomized to no expert panel review, they will discuss with their surgeon the best surgical option for them and proceed as they would in standard of care. Patients with symptomatic lumbar spinal stenosis and single level degenerative grade I spondylolisthesis will be treated either with decompression or decompression with fusion. Symptomatic spinal stenosis will be defined as radicular and/or back pain either induced by or aggravated by activity and relieved by rest in a patient with either moderately severe or severe lumbar spinal stenosis. Patient-reported outcomes will be captured at baseline, at 3 and 6 months, and annually out to five years.

The imaging data will be used to create artificial intelligence (AI) algorithms that will help assess when an expert panel is more likely to suggest one treatment over the other as well as develop an algorithm that would prospectively classify patients as either 'stable' or 'unstable.' Ultimately long term follow-up will help confirm whether a case was correctly assessed as stable or unstable. A patient would be confirmed as unstable, if they underwent decompression alone and then required a re-operation to stabilize the spine at the level of spondylolisthesis within 5 years of the initial operation. In a similar way, a patient would be confirmed as stable, if no re-operation were necessary over the 5-year study follow-up period.

Select sites will participate in an assessment of the utilization of step count as an outcome. Average step count will be captured pre-operatively as well as at 3- and 6-months and annually out to 5 years. The mean step count at each time point will be compared to the mean change scores for ODI and EQ-5D. Additionally, average step counts overtime will be analyzed for those patients who undergo a re-operation.

Interim Analysis: An interim analysis is planned when 150 patients have reached eligibility at 6 month follow-up. Patients' change from baseline patient-reported outcome questionnaires will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic lumbar spinal stenosis: defined as radicular and/or back pain either induced or aggravated by activity and relieved by rest.
* Single-level grade I degenerative spondylolisthesis (3-14mm)

Exclusion Criteria:

* Serious medical illness (ASA Class IV or higher)
* Spondylolysis
* Multilevel spondylolisthesis or high grade spondylolisthesis (grade II or greater than 14mm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 662 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
EuroQol-5 Dimensions (EQ-5D) | 1 year, 2 years, 3 years, 4 years, 5 years
  Quality of life will be assessed through EuroQol 5 Dimensions (EQ-5D) at all time points. Analysis will focus on mean change score as well as the percentage of patients who fail to improve EQ-5D score at each time point. Patients randomized to expert panel review will be compared to those without expert panel review.
NASS patient satisfaction scale | 1 year, 2 years, 3 years, 4 years, 5 years
  The percentage of patients who achieve NASS patient satisfaction score of 1 or 2 will be compared at each time point between those patients who were randomized to an expert panel review or not.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Baseline, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  To determine at 1 and 2 years if an expert panel review of individual cases is associated with a greater percentage of patients who improve by more than 10 points. In addition, we will compare mean change in ODI score among patients randomized to expert panel review to those randomized to receive no review.
Oswestry Disability Index (ODI) | Baseline, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  To compare mean change in ODI score between patients treated with laminectomy alone versus laminectomy with instrumented lumbar fusion
EuroQol-5 Dimensions (EQ-5D) | Baseline, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Quality of life will be assessed through EuroQol 5 Dimensions (EQ-5D) at all time points. The three-level scale denotes no problems, some problems, or extreme problems, across the five domains of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. A visual analog scale is also used to evaluate overall health state. Comparisons among groups will compare difference in the change scores.
Cost Data -- Hospital Claims & Health Resource Utilization | 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Costs will also be compared between groups during the duration of the study.
Complications | 1 month
  Complications at time of surgery to 30 days post-operative will be collected.
Return to Work | Baseline, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Working status will be asked at all time points to capture productivity.
Flexion-Extension Radiographs | Baseline, 1 year, 2 years
  To determine stability after surgery as well as fusion.
36-inch Standing Plain Radiographs | Baseline, 1 year
  To assess spine alignment.

CONTACTS AND LOCATIONS:
Overall Officials: Zoher Ghogawala, MD, Principal Investigator — Lahey Hospital & Medical Center
Locations (17):
- United States (16):
  - Barrow Brain and Spine, Scottsdale, Arizona
  - University of California, San Fransisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Carle Neurosciences Institute, Urbana, Illinois
  - Goodman Campbell Brain & Spine, Carmel, Indiana
  - Norton Leatherman Spine Center, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Hospital for Special Surgery, New York, New York
  - Columbia University, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah Hospital, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin
- University Health Network - Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data would be shared with other researchers after primary analysis has been published.
Supporting Information: Study Protocol, SAP
Time Frame: After primary analysis has been published for up to 5 years.

REFERENCES:
- [Derived] Ghogawala Z, Rizvi TZ, Lin Z, Kanter A, Mummaneni PV, Bisson EF, Albert TJ, Resnick DK, Wang MY, Glassman S, Polly DW Jr, Bydon M, Magge SN, Tumialan LM, Fehlings MG, Steinmetz MP, Whitmore RG, Rajshekhar V, Harrop JS, Hartl R, Ahmed E, Coric D, McCormick PC, Assaker R, Msaddi AK, Holly LT, Kawaguchi Y, Falavigna A, Barker FG 2nd, Benzel EC; SLIP II Investigators. Use of an Expert Panel for Symptomatic Patients With Grade I Degenerative Lumbar Spondylolisthesis: A Randomized Clinical Trial. Neurosurgery. 2025 Nov 6. doi: 10.1227/neu.0000000000003838. Online ahead of print. PMID 41196064